CLINICAL TRIAL: NCT07097298
Title: Empathy and (Self-)Compassion to Improve the Quality of Life of Parkinson's Disease Patients and Caregivers: an Exploratory Study
Brief Title: Empathy and (Self-)Compassion in Parkinson's Disease Patients and Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alain Kaelin (Other)
Collaborators: CTU-EOC Clinical Trial Unit Ente Ospedaliero Cantonale (Unknown)
Responsible Party: Sponsor-Investigator, Alain Kaelin, Prof. MD PhD, Ente Ospedaliero Cantonale, Bellinzona
Organization: Ente Ospedaliero Cantonale, Bellinzona (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: EMPCOMP-PD-001
Record Dates: First submitted 2025-07-17; First posted 2025-07-31 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Parkinson Disease(PD)
Keywords: Empathy; (self-)compassion; Parkinson disease (PD)
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Empathy and (self-)compassion training (Experimental): A 6-week empathy and compassion training will be designed and delivered involving PD patients and caregivers. During the compassion training participants will do mindfulness, writing and poetry exercises addressing the cognitive, emotional, motivational and behavioural components of (self-)compassion. The training will be designed in order to address both self-compassion and compassion. We expect to conduct 1 session at the beginning and 1 session at the end of the program with exercises to do at home for 6 weeks, assigned as tasks based on the needs of patients and their caregivers
  Interventions: Behavioral: empathy and compassion training

INTERVENTIONS:
Behavioral: empathy and compassion training — A 6-week empathy and compassion training will be designed and delivered involving PD patients and caregivers. During the compassion training participants will do mindfulness, writing and poetry exercises

SUMMARY:
The goal of this clinical trial is to improve quality of life in Parkinson's Disease (PD) patients by increasing their empathy and their (self-)compassion. The main question it aims to answer is:

Does the level of quality of life in PD patients and caregivers improve after empathy/(self-)compassion training?

Participants will be delivered a 6-week empathy and compassion training (mindfulness, writing and poetry exercises addressing the cognitive, emotional, motivational and behavioural components of (self-)compassion) and will also be asked to answer questionnaires before and after the training

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PD
* Hoehn and Yahr scale, stage ≤ 3
* Mini Mental State Examination with a score ≥ 26
* Able to give informed consent as documented by signature
* At least, secondary school education
* To have a regular caregiver at home

Exclusion Criteria:

* Any medical condition that is not PD, such as drug induced parkinsonism
* Major depression, dysthymia, or according to DSM-V
* Other neurological or psychiatric diseases
* Neuropsychological scores compatible with the diagnosis of early dementia
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, etc

For CAREGIVERS:

Inclusion criteria

* Taking care of the patient on a regular basis, i.e., at least 3 days per week
* Being caregiver of the patients for at least 3 months
* At least, secondary school education
* Written informed consent

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
PD patients quality of life improvement | from baseline to the end of intervention (6weeks)
  the change (no min / max values foreseen) in the level of quality of life in PD patients as measured by the Parkinson's Disease Questionnaire (PDQ-8), which assesses 8 domains of quality of life: mobility, activities of daily of living, emotional well-being, stigma, social support, cognition, communication, and bodily discomfort; higher scores indicate a worse quality of life

SECONDARY OUTCOMES:
change in the level of empathy in PD patients and caregivers | from baseline to the end of intervention (6weeks)
  change in the level of empathy in PD patients and caregivers as measured by Interpersonal Reactivity Index (IRI): this questionnaire captures both the cognitive and emotional facets of empathy. It includes four seven-item subscales: 1) Fantasy (F) and 2) Perspective Taking (PT) for the cognitive dimension and 3) Empathic Concern (EC) and 4) Personal Distress (PersDis) for an emotional one. The F scale assesses the tendency to identify oneself imaginatively in characters and situations (for example, movie characters and novels); the PT scale contains elements that map to the ability to apply the perspectives of other people from their point of view; the EC scale evaluates feelings of compassion and concern regarding other people; the PersDis measures the personal feelings of anxiety and discomfort that are experienced by observing the negative emotion
self-compassion level change in PD patients and caregivers | from baseline to the end of intervention (6weeks)
  change in the level of self-compassion in PD patients and caregivers as measured by Self-Compassion Scale (SCS): this is a 26-item validated questionnaire which measures self-compassion with six subscales: self-kindness, self-judgment, common humanity, isolation, mindfulness, and over-identification. Past studies used this test with people with Parkinson's . The total self-compassion score is the mean of the six subscale means and ranges from 1 to 5, with a higher score indicating greater self-compassion
compassion level change in PD patients and caregivers | from baseline to the end of intervention (6weeks)
  change in the level of compassion in PD patients and caregivers as a derived measure of the SCS: a 26-item validated questionnaire, measures self-compassion with six subscales: self-kindness, self-judgment, common humanity, isolation, mindfulness, and over-identification. Past studies used this test with people with Parkinson's. The total self-compassion score is the mean of the six subscale means and ranges from 1 to 5, with a higher score indicating greater self-compassion
quality of life level change in caregivers | from baseline to the end of intervention (6weeks)
  change in the level of quality of life in caregivers as measured by the Family Caregiver Quality of Life Scale (FAMQOL): it evaluates caregivers' quality of life across multiple dimensions (physical, psychological, and social well-being). The FAMQOL consists of 16 self-reported questions with 5-option Likert responses, ranging from "Strongly Disagree" to "Strongly Agree"

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto di Neuroscienze Cliniche della Svizzera Italiana, EOC, Lugano, Switzerland